CLINICAL TRIAL: NCT04240132
Title: Relation Between Adherence to Hand Hygiene Practices by Healthcare Providers Working in Intensive Care Unit and Microbial Contamination on Feeding Tubes and Other Components of Feeding Systems
Brief Title: Hand Hygiene Practices and Microbial Contamination on Feeding Tubes and Other Components of Feeding Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Collaborators: Turkish Society of Clinical Enteral and Parenteral Nutrition (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Assistant Professor, Istanbul Demiroglu Bilim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01/2020
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Enteral Nutrition; Microbial Colonization; Adherence
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, observational and semi-experimental (mix method)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adherence to hand hygene (Experimental): The face-to-face interview will be held in an appropriate empty room in the intensive care unit (ICU) in a time schedule suitable for the healthcare workers. The researchers will provide training to healthcare workers working in the ICU in accordance with the World Helath Organization (WHO) Hand Hygiene Guidelines. One day training on nursing interventions related to enteral feeding treatment will be provided to nurses and their questions will be answered. At the end of the each training, trainees will be given a data collection form to assess the effectiveness of the training.
  Interventions: Other: Adherence to Hand Hygiene

INTERVENTIONS:
Other: Adherence to Hand Hygiene — determine the colonization of microorganisms due to microbial reproduction on the external surface of the distal end of the enteral feeding tube (EFT), hub of the EFT and other feeding system components and assess the relation between the colonization and adherence to hand hygiene practices by nurses and other healthcare workers

SUMMARY:
Enteral feeding tube (EFT) and component of feeding systems can serve as a reservoir of microorganisms, and the main reason is inappropriate hand hygiene practices. The aim of the project is to determine colonization of microorganisms on the EFT and other components and assess the relation between colonization and adherence to hand hygiene practices by healthcare workers in the intensive care unit.

This prospective, observational and semi-experimental study will be conducted in one year. The project will be completed with healthcare workers and 51 patients who are feeding enteral route via nasogastric tube at least for three days. The researchers will provide training to healthcare workers in accordance with the World Health Organization (WHO) Hand Hygiene Guidelines. Hand hygiene behaviors of the participants will be observed and the question forms will be filled before and after training by researchers. The samples for microbial analysis will be collected from the EFT by sterile swaps.

DETAILED DESCRIPTION:
Enteral Feeding Tube (EFT) such as Nasogastric Tube (NGT), Duodenal/Jejunal Tube and Gastrostomy Tube are frequently used in Intensive Care Unit (ICU). However, EFT is generally an omitted/neglected source of contamination. EFT can serve as a reservoir of Methicillin Resistant Staphylococcus Aureus (MRSA), which multiplies the risk of mortality by 2-2.5 times, for microorganism transmission. As a consequence of contamination of EFT, microorganisms, that may be manifest with the symptoms such as abdominal pain, distention, nausea, vomiting, diarrhea, may reproduce and progress to bacteremia, septicemia and even to death. In some studies, it is observed that there is a relation between the contamination on the external surface of EFT and contamination on the entry of EFT (hub), and it is also reported that the rate of contamination on the hub of the EFT and the environment of the patient is quite high. ICU nurses are responsible for sustaining safe and secure feeding, medication and fluid replacement of patients. Also, they provide enteral feeding products to patients as they are prescribed. Personnel training, proper processing procedures and developed enteral feeding protocols are shown to decrease the incidence of bacterial contamination on the enteral feeding tube

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years old or older
* Being enteral fed via nasogastric tube at least for three days
* Patients' relatives approve to be enrolled are going to be included in the study
* Nurses and other healthcare providers who work in the ICU

Exclusion Criteria:

* Patients who are being under respiratory, contact or droplet isolation according to definitions of Centers for Disease Control and Prevention
* Patients' relatives do not approve enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Adherence to hand hygiene at nurses | up to 12 weeks
  Hand Hygiene Belief Scale will be used. The scale consists of 22 items on individual's beliefs on hand hygiene and perceptions on the importance of hand hygiene. The lowest total score is 22 and the highest total score is 110. Higher scores can be interpreted as having positive beliefs on hand hygiene.
Adherence to hand hygiene at auxillary service staff | up to 12 weeks
  Scale for Hand Hygiene Compliance of Auxillary Service Staff will be used. It consist of 21 items and has 4 dimensions; "After contact with patient" (6 items), "Before contact with patient" (6 items), "risk of contact with blood and body fluids" (4 items), "after contact with patient environment" (5 items). The lowest total score is 0 and the highest total score is 84. Higher scores represent higher adherence to hand hygiene.
Microbial contamination rate | up to 12 weeks
  The samples for microbial analysis will be collected from internal and external surface of the NGT and other components of the feeding system by sterile swaps from all of the participant patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Ozen, Principal Investigator — Demiroglu Bilim Üniversitesi
Locations (1):
- Demiroglu Bİlim University, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhalla A, Pultz NJ, Gries DM, Ray AJ, Eckstein EC, Aron DC, Donskey CJ. Acquisition of nosocomial pathogens on hands after contact with environmental surfaces near hospitalized patients. Infect Control Hosp Epidemiol. 2004 Feb;25(2):164-7. doi: 10.1086/502369. PMID 14994944
- [Result] Duckro AN, Blom DW, Lyle EA, Weinstein RA, Hayden MK. Transfer of vancomycin-resistant enterococci via health care worker hands. Arch Intern Med. 2005 Feb 14;165(3):302-7. doi: 10.1001/archinte.165.3.302. PMID 15710793
- [Result] Ho SS, Tse MM, Boost MV. Effect of an infection control programme on bacterial contamination of enteral feed in nursing homes. J Hosp Infect. 2012 Sep;82(1):49-55. doi: 10.1016/j.jhin.2012.05.002. Epub 2012 Jul 4. PMID 22765960
- [Result] Mathus-Vliegen EM, Bredius MW, Binnekade JM. Analysis of sites of bacterial contamination in an enteral feeding system. JPEN J Parenter Enteral Nutr. 2006 Nov-Dec;30(6):519-25. doi: 10.1177/0148607106030006519. PMID 17047178